CLINICAL TRIAL: NCT02202018
Title: Patient and Provider Education for Patients With Severe Chronic Kidney Disease: Assessing the Impact on Barriers and Use of Home Dialysis
Brief Title: A Cluster Randomized Trial to Assess the Impact of Patient and Provider Education on Use of Home Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Braden Manns, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REB13-0083_MOD1
Record Dates: First submitted 2014-07-11; First posted 2014-07-28 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Disease
Keywords: Knowledge Translation; Chronic Kidney Disease; Dialysis; Home dialysis; Cluster randomized trial
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active KT Intervention (Experimental): CKD clinics receiving the active knowledge translation intervention.
  Interventions: Other: Active KT intervention
- Usual standard of care (No Intervention): Clinics will continue their standard of care education and approach to use of home dialysis.

INTERVENTIONS:
Other: Active KT intervention — 1. Provider & patient-directed infographics educating patients about home dialysis will be displayed in prominent clinic wall space
  2. Educational white board presentations promoting home dialysis
  3. Each clinic will receive reports outlining their current use of home dialysis in incident ESRD patients compared with provincial & national averages
  4. A Canadian version of the MATCH D tool will be provided to clinic staff, to help evaluate patient appropriateness for home dialysis.
  5. Each clinic will receive an in-person visit from one of the study investigators/collaborators detailing the benefits of home dialysis, and the educational tools being offered to support care within their clinic.
  Arms: Active KT Intervention

SUMMARY:
Patients with severe kidney failure require dialysis or transplantation to survive. For those in whom a transplant is not an option, there are two main dialysis options: hemodialysis (either incenter or at home) or home peritoneal dialysis. Home-based therapies (peritoneal and home hemodialysis) are under-utilized in many Canadian jurisdictions with the proportion of home-based therapies varying between 10 and 40% across centres. Studies show that the low use of home dialysis is due to a variety of factors, though patient and provider awareness and knowledge of home dialysis are major factors. In this cluster randomized trial, the investigators will determine whether a standardized modality education program directed at patients, in combination with a provider-directed intervention, can increase the use of home dialysis in incident dialysis patients in Canada.

DETAILED DESCRIPTION:
Background: Patients with severe kidney failure require dialysis or transplantation to survive. For those in whom a transplant is not an option, there are two main dialysis options: hemodialysis (either incenter or at home) or home peritoneal dialysis. Home-based therapies (peritoneal and home hemodialysis) are under-utilized in many Canadian jurisdictions with the proportion of home-based therapies varying between 10 and 40% across centres. The use of home dialysis remains lower than expected due to combination of patient, caregiver, provider, and health system barriers. Previous studies have highlighted several potential patient and caregiver barriers to use of home therapies including knowledge, skills, personal circumstances, and social supports. Provider barriers have been reported to include lack of training in peritoneal dialysis, lack (or perceived lack) in skills and knowledge, bias, and possibly inadequate physician reimbursement for home dialysis.

The Canadian Kidney Knowledge Translation and Generation Network (CANN-NET), a national network of clinicians, researchers and knowledge users that was established to ensure best practices for patients with chronic kidney disease (CKD), recently created dialysis modality educational tools aimed at patients and kidney health care providers. On behalf of CANN-NET, the investigators propose a cluster randomized controlled trial (with clusters consisting of severe CKD clinics) of a knowledge translation (KT) strategy to increase use of home dialysis in patients with end-stage renal disease. Informed by careful survey work, clinics randomized to the knowledge translation intervention will receive patient and provider directed educational tools, including the MATCH D tool, compelling visual aids (infographic, white board animated video, and an educational video on dialysis modality options), audit and feedback, and in-person medical detailing. Control clinics will continue with their usual practice with respect to dialysis modality education.

Primary Objective To determine whether a standardized modality education program directed at patients, in combination with provider-directed interventions can increase the use of home dialysis in incident dialysis patients in Canada

Study Design: A cluster randomized trial of CKD clinics across Canada comparing the efficacy and safety of a KT intervention aiming to increase use of home dialysis in patients with advanced CKD. The unit of observation will be the patient (i.e., outcomes will be measured at the level of an individual patient), and the unit of randomization will be at the level of the multidisciplinary CKD clinic.

Team: The investigative study team includes experts in the clinical epidemiology of CKD and kidney failure, local opinion leaders from every province/region, as well experts in knowledge translation and cluster randomized design. As such, the investigators are well positioned to carry out the proposed study.

Research Significance: Home dialysis, in comparison to incenter hemodialysis, is associated with increased patient independence, better clinical outcomes, and lower health care costs. Due to a variety of factors, home dialysis use remains variable across Canada. This study will test the effectiveness of a KT strategy to increase the use of home dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Multidisciplinary clinics in Canada that provide care coordinated by a Nephrologist to patients with chronic kidney disease (CKD). These clinics have already been identified in a previous survey

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Outcome: Use of home dialysis | Use of home dialysis at six months after dialysis initiation
  Proportion of patients with incident end-stage renal disease initiating dialysis after the intervention who are using home dialysis (home hemodialysis or peritoneal dialysis) six months after dialysis initiation. Use of home dialysis will be ascertained from the clinic clusters and confirmed by linkage with the Canadian Organ Replacement Register (CORR).

SECONDARY OUTCOMES:
Secondary outcome: Use of home dialysis at six months in patients who have been followed by a Nephrologist | Use of home dialysis at six months after dialysis initiation in patients who have been followed by a Nephrologist
  Proportion of patients with incident end-stage renal disease initiating dialysis after the intervention who were followed by a Nephrologist prior to dialysis initiation who are using home dialysis (home hemodialysis or peritoneal dialysis) six months after dialysis initiation. Use of home dialysis will be ascertained from the clinic clusters and confirmed by linkage with the Canadian Organ Replacement Register (CORR).

CONTACTS AND LOCATIONS:
Overall Officials: Navdeep Tangri, MD PhD FRCPC, Study Director — University of Manitoba; Braden Manns, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Derived] Manns BJ, Garg AX, Sood MM, Ferguson T, Kim SJ, Naimark D, Nesrallah GE, Soroka SD, Beaulieu M, Dixon SN, Alam A, Allu S, Tangri N. Multifaceted Intervention to Increase the Use of Home Dialysis: A Cluster Randomized Controlled Trial. Clin J Am Soc Nephrol. 2022 Apr;17(4):535-545. doi: 10.2215/CJN.13191021. Epub 2022 Mar 21. PMID 35314481